CLINICAL TRIAL: NCT02238730
Title: Comparative Efficacy and Cognitive Side-Effects of Ultrabrief Right Unilateral Electroconvulsive Therapy and Brief Pulse Bitemporal Electroconvulsive Therapy
Brief Title: Ultrabrief Right Unilateral and Brief Pulse Bitemporal Electroconvulsive Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Resources not available for the study
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KPSC IRB10133; KPSC IRB 10133 (Other: Kaiser Permanente Southern California IRB)
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Depression; Depressive Disorder; Treatment Resistant Depressive Disorder; Bipolar Disorder; Major Depressive Disorder
Keywords: Depression; Depressive Disorder; Treatment Resistant Depressive Disorder; Bipolar Disorder; Major Depressive Disorder; Electroconvulsive therapy
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Treatment-Resistant; Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrabrief Right Unilateral (Active Comparator): Ultrabrief (0.25 ms) Right Unilateral Electroconvulsive Therapy
  Interventions: Device: Ultrabrief Right Unilateral
- Brief Pulse Bitemporal (Active Comparator): Brief Pulse (0.5 ms) Bitemporal Electroconvulsive Therapy
  Interventions: Device: Brief Pulse Bitemporal

INTERVENTIONS:
Device: Ultrabrief Right Unilateral — The first six electroconvulsive therapy sessions using ultrabrief (0.25 ms) right unilateral electroconvulsive therapy
  Other Names: Thymatron System IV
  Arms: Ultrabrief Right Unilateral
Device: Brief Pulse Bitemporal — The first six electroconvulsive therapy sessions using brief pulse (0.5 ms) bitemporal electroconvulsive therapy
  Other Names: Thymatron System IV
  Arms: Brief Pulse Bitemporal

SUMMARY:
To evaluate the equivalent efficacy of ultrabrief pulsewidth right unilateral electroconvulsive therapy versus bitemporal brief pulse electroconvulsive therapy in the treatment of depression and to evaluate the cognitive effects of ultrabrief right unilateral electroconvulsive therapy versus bitemporal brief pulse electroconvulsive therapy.

DETAILED DESCRIPTION:
Patients will be randomized to either bitemporal brief pulse electroconvulsive therapy ( 0.5 ms pulse width) or right unilateral ultrabrief pulse electroconvulsive therapy for the first six treatments. If further treatment is necessary, electrode placement will be chosen by the treating psychiatrist. All electroconvulsive therapy treatments will be performed with a Thymatron System IV instrument. (Somatics, LLC, Lake Bluff, Illinois, USA) Pre- electroconvulsive therapy testing will occur within one week of beginning treatment. Post-electroconvulsive therapy testing will occur within 48 hours of the 6th treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients age 18 and above referred for electroconvulsive therapy will be screened for eligibility for participation in this study.
* Basic competency in English
* Diagnosis of either of the following:

  1. Major Depressive Disorder, Single Episode
  2. Major Depressive Disorder, Recurrent
  3. Bipolar Disorder, Currently Depressed

Exclusion Criteria:

* Pre-existing cognitive impairment with an initial Mini Mental Status Exam Score of 24 or lower
* Major neurological disease
* Other medical conditions making electroconvulsive therapy an excessive risk to be completed safely in an outpatient surgery center and anticonvulsant therapy.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HAMD) | up to 2-3 weeks
  Standardized assessment administered by a psychologist

SECONDARY OUTCOMES:
Mini Mental Status Examination | up to 2-3 weeks
  Standardized assessment administered by a psychologist

CONTACTS AND LOCATIONS:
Overall Officials: Ronad L Warnell, MD, Principal Investigator — Kaiser Permanente